CLINICAL TRIAL: NCT05125003
Title: Parent-implemented Treatment for Repetitive Behaviors in Children With ASD: Using a Novel Telehealth Approach to Increase Service Access.
Brief Title: Family-Implemented Treatment on the Behavioral Inflexibility of Children With Autism
Acronym: FITBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD105036 (NIH)
Record Dates: First submitted 2021-10-29; First posted 2021-11-18 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Autism Spectrum Disorder; Repetitive Compulsive Behavior
Keywords: family-based intervention; video-conferencing technology; telehealth
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FITBI (Experimental): Reinforcement-based learning procedures delivered via telehealth in 16 remote-delivered treatment sessions - 13 weekly and 3 booster treatment sessions over 6 month period.
  Interventions: Behavioral: FITBI
- Parent Education (Active Comparator): Information relevant to parenting a young child with ASD (e.g. parent advocacy, developmental changes in ASD, treatment options) delivered via telehealth in 15 remote-delivered treatment sessions -12 weekly and 3 booster treatment sessions over 6 month period.
  Interventions: Behavioral: Parental Education

INTERVENTIONS:
Behavioral: FITBI — parents learn to identify high probability cues in the environment that can elicit RRBI symptoms and teach their child to inhibit repetitive behaviors and instead replace them with alternative and flexible play behaviors; and (b) teach parents how to embed this FITBI approach into their child's everyday routines
  Arms: FITBI
Behavioral: Parental Education — Sessions will cover relevant information on young children with ASD, including understanding the ASD diagnosis, developmental changes in ASD, educational planning, advocacy, and treatment options.
  Arms: Parent Education

SUMMARY:
The overall goal of this project is to determine whether a new form of family-based treatment for repetitive and inflexible behaviors, delivered using videoconferencing technology, can counter any negative effects of those behaviors, but also improve positive outcomes for young children with ASD.

DETAILED DESCRIPTION:
The overall goal of this project is to conduct a parallel group randomized controlled trial comparing remote delivery of FITBI (13-week intervention + 3 booster sessions over 6 months) to remote delivery of a parent education only (PE) control condition in a final sample size of 100 (3 years, 0 months to 9 years, 6 months) children with ASD and high rates of ritualistic repetitive behaviors. We will use TORSH, a comprehensive secure online platform that enhances therapist-parent coaching via telehealth. Further, an important objective of this proposal is to examine child and parent factors associated with treatment response and uptake in order to advance translational research and knowledge on personalized intervention approaches. Thus, the aims of this project are to:

Aim 1: Examine the acute and distal effects of the FITBI intervention on child and parent outcomes.

H1: In comparison to a PE only condition, FITBI will result in reductions in children's repetitive behaviors and increases in appropriate play skills immediately post-treatment.

H2: Effects of the FITBI intervention will be maintained at a 6-month follow-up and increases in child adaptive functioning and decreases in parent stress will be found.

Aim 2: Determine if the FITBI intervention shows differential treatment effects for lower versus higher order repetitive behaviors.

H1: FITBI will be effective at treating both lower and higher order RRBIs.

Aim 3: Examine if child variables (i.e., IQ and anxiety) moderate treatment response.

H1: Based on prior behavioral intervention research, it is hypothesized that children with higher IQs and fewer symptoms of anxiety at pretreatment, will show a better treatment response.

Aim 4: Explore if parent variables (i.e., SES, race/ethnicity, marital status, and stress) predict intervention fidelity and telehealth acceptance.

H1: As this is an exploratory aim, we do not have specific hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* ASD criteria on Social Communication Questionnaire-Lifetime and Autism Diagnostic Interview-Revised.
* Between ages of 3 years, 0 months and 9 years, 6 months
* exhibiting clinically significant levels of repetitive behavior (Score >26 on Repetitive Behavior Scales-Revised
* prior clinical or medical diagnosis of autism spectrum disorder

Exclusion Criteria:

* diagnosed comorbid genetic disorder known to associated with increased symptom severity
* child engages in serious self-injurious behavior with intensity or frequency that warrants hospitalization
* change in psychotropic medications within last 6 weeks
* child already receives >20hours per week of home-based ABA services

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Behavioral Inflexibility Scale - Clinical Interview | Baseline
  video interview yields a severity score from 0 no impairment to 28 maximum impairment
Behavioral Inflexibility Scale - Clinical Interview | 6 weeks
  video interview yields a severity score from 0 no impairment to 28 maximum impairment
Behavioral Inflexibility Scale - Clinical Interview | 12 weeks
  video interview yields a severity score from 0 no impairment to 28 maximum impairment
Behavioral Inflexibility Scale - Clinical Interview | 6 months
  video interview yields a severity score from 0 no impairment to 28 maximum impairment

SECONDARY OUTCOMES:
Aberrant Behavior Checklist-Community (ABC-C) | Baseline, 6 weeks, 12 weeks, and 6 month follow-up
  online survey
Direct Observation of Repetitive Behaviors in Autism (DORBA) | Baseline, 12 weeks, and 6 month follow-up
  The DORBA is an observational measure of restricted and repetitive behaviors in children with ASD based on clinician- or caregiver-child interactions.
Behavioral Inflexibility Scale (BIS) | Baseline, 6 weeks, 12 weeks, and 6 month follow-up
  parent survey of severity with total score ranging from 0 (no problem) to 190 very severe on all 38 items

CONTACTS AND LOCATIONS:
Overall Officials: Brian Boyd, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Juniper Gardens Children's Project, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant data will be shared with the NDAR repository using their system of GUIDs.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available following the completion of the trial and data cleaning. It will remain in the archive as soon as the archive is supported.
Access Criteria: Access criteria will be managed by the NDAR site.